CLINICAL TRIAL: NCT04090736
Title: A Randomized Phase III, Multicentre, Open Label Clinical Trial Comparing Azacitidine Plus Pevonedistat Versus Azacitidine in Older/Unfit Patients With Newly Diagnosed Acute Myeloid Leukemia Who Are Ineligible for Standard Induction Chemotherapy
Brief Title: Study to Compare Azacitidine Plus Pevonedistat Versus Azacitidine in Patients With Acute Myeloid Leukemia Not Eligible for Standard Chemotherapy
Acronym: PEVOLAM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Dynamic Science S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEVOLAM
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Leukemia; Myeloid; Acute; Pevonedistat; Azacitidine; Randomized; Clinical trial
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — pevonedistat; Azacitidine

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, multicenter, open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Pevonedistat plus Azacitidine (Experimental): Pevonedistat 20 mg/m2 IV on days 1, 3, and 5 plus Azacitidine 75 mg/m2 subcutaneous administered on a 5-on/2-off [weekend]/2-on schedule in 28-day cycles (intravenous Azacitidine can be administered for any patients who have non-tolerated local reactions)
  Interventions: Drug: Pevonedistat; Drug: Azacitidine
- Arm B: Azacitidine (Active Comparator): Azacitidine 75 mg/m2 subcutaneous on a 5-on/2-off [weekend]/2-on schedule in 28-day cycle (intravenous azacitidine can be administered for any patients who have non-tolerated local reactions)
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Pevonedistat — Pevonedistat 20 mg/m2 intravenous on days 1, 3, and 5 (28-day cycles)
  Arms: Arm A: Pevonedistat plus Azacitidine
Drug: Azacitidine — Azacitidine 75 mg/m2 subcutaneous on a 5-on/2-off [weekend]/2-on schedule (28-day cycle). Intravenous for patients who have non-tolerated local reactions

SUMMARY:
Randomized phase III, multicentre, open label clinical trial to compare pevonedistat in combination with azacytidine versus azacytidine alone, which can be considered a standard of care for patients with newly diagnosed acute myeloid leukemia not eligible for intensive chemotherapy (thus not eligible for an allogeneic hematopoietic stem cell transplant.

DETAILED DESCRIPTION:
Prospective, 1:1 randomized multicentre, open label, phase III clinical trial to evaluate efficacy and safety of pevonedistat in combination with azacytidine versus azacytidine in the treatment of naïve adult patients with acute myeloid leukemia who are not eligible for standard induction therapy due to age, co-morbidities or risk-factors.

Subjects will be randomized to one of the two treatment arms in a 1:1 ratio, both of which will have treatment cycles of 28 days:

* Arm A: Pevonedistat (PEVO) 20 mg/m2 IV on days 1, 3, and 5 plus Azacitidine (AZA) 75 mg/m2 subcutaneous (SC) administered on a 5-on/2-off [weekend]/2-on schedule in 28-day cycles (IV AZA can be administered for any patients who have non-tolerated local reactions)
* Arm B: AZA 75 mg/m2 SC on a 5-on/2-off [weekend]/2-on schedule in 28-day cycle (IV AZA can be administered for any patients who have non-tolerated local reactions)

  466 subjects will be randomized in the study. Subjects will continue their study treatment until documented disease progression per Investigator assessment, unacceptable toxicity, withdrawal of consent, or the subject meets other protocol criteria for discontinuation

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or older
2. Morphological diagnosis of Acute Myeloid Leukemia (AML) (WHO criteria 2008)
3. Subject must have an Eastern Cooperative Oncology Group (ECOG) Performance status (PS) of 0 to 3 (ECOG 0-2 for patients greater than or equal to 75 years old).
4. Newly diagnosed AML
5. Patient must be considered be ineligible for treatment with a standard Ara-C and anthracycline induction regimen due to age or co-morbidities defined by one of the following:

   1. ≥ 75 years of age
   2. Or ≥ 18 to 74 years of age with at least one of the following:

      * ECOG Performance Status of 2 or 3;
      * Cardiac history of cardiac heart failure requiring treatment or Ejection Fraction ≤ 50% or chronic stable angina;
      * Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) ≤ 65% or Forced Expiratory Volume in 1 second (FEV1) ≤ 65% or significant history of chronic pulmonary obstructive disease;
      * Glomerular filtration rate (GFR) ≥ 30 mL/min to < 50 ml/min or levels of creatinine between the upper limit of the normal range (ULN) and 2.5 mg/dL (≤ 250 μmol/l).
      * Hepatic impairment with total bilirubin > 1.5 to ≤ 3 × ULN or with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2.5×ULN to ≤ 5×ULN
      * Non active/controlled prior neoplastic disease
      * Any other patient´s comorbidity or disease condition that the physician judges to be incompatible with intensive chemotherapy must be reviewed, documented, and approved by the Sponsor before study enrollment).
6. Clinical laboratory values within the following parameters (repeat within 3 days before the first dose of study drug if laboratory values used for randomization were obtained more than 3 days before the first dose of study drug):

   * Total bilirubin ≤ 1.5 × ULN except in patients with Gilbert's syndrome or ≤ 3 × ULN if elevation is attributed to underlying leukemia. Patients with Gilbert's syndrome may enroll with direct bilirubin ≤3 × ULN of the direct bilirubin. Elevated indirect bilirubin due to posttransfusion hemolysis is allowed.
   * ALT and AST ≤ 2.5×ULN or ≤ 5×ULN if elevation is attributed to underlying leukemia.
   * Adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min (calculated by the Cockcroft Gault formula, (see Appendix 5).
   * Albumin >2.7 g/dL.
7. Subject has a white blood cell count <50 × 109/L. Patients who are cytoreduced with leukapheresis or with hydroxyurea may be enrolled if they meet the eligibility criteria before starting therapy.
8. Female subjects must be either postmenopausal for at least 1 year before screening (see Appendix 12 for definition) OR permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy) OR Women of Childbearing Potential (WOCBP) must agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception (see Appendix 11), at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), or Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception). Female subjects of childbearing potential must have negative results for pregnancy test performed and must not be lactating and breastfeeding.
9. Male subjects even if surgically sterilized (i.e., status post vasectomy), who are sexually active, must agree, from Study Day 1 through at least 4 months after the last dose of study drug, to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
10. Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Previous treatment for myelodysplastic síndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML) or myeloproliferative neoplasms (MPN), with chemotherapy or other antineoplastic agents including HMAs (up to 2 cycles of Hypomethylating agents (HMA) such as decitabine or azacitidine. Previous treatment is permitted with hydroxyurea and with lenalidomide, except that lenalidomide may not be given within 8 weeks before the first dose of study drug.
2. Subject has history MPN with BCR-ABL1 translocation and AML with BCR-ABL1 translocation.
3. Genetic diagnosis of acute promyelocytic leukemia.
4. Eligible for intensive chemotherapy and/or allogeneic stem cell transplantation.

   * The reason a patient is not eligible for intensive chemotherapy and/or allogeneic stem cell transplantation is described in the inclusion criteria section
   * The reason a patient is not eligible for intensive chemotherapy must be documented in the electronic case report form (eCRF).
5. Patients with either clinical evidence of or history of central nervous system involvement by AML.
6. Diagnosed or treated for another malignancy within 1 year before randomization or previously diagnosed with another malignancy and have any evidence of residual disease which may compromise the administration of AZA or AZA+PEVO.
7. Psychological,social, or geographic factors that otherwise preclude the patient from giving informed consent, following the protocol, or potentially hamper compliance with study treatment and follow-up.
8. Subject has a white blood cell count > 50 × 109/L.
9. Contraindications for PEVO or AZA.
10. Known hypersensitivity to pevonedistat or its excipients.
11. Female patients who intend to donate eggs (ova) during the course of this study or for 4 months after receiving their last dose of study drug(s).
12. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
13. Male patients who intend to donate sperm or father a child during the course of this study or for 4 months after receiving their last dose of study drug(s).
14. Subject is known to be positive for HIV (HIV testing is not required for eligibility assessment). Known HIV positive patients who meet the following criteria will be considered eligible:

    * Cluster of differentiation 4 (CD4) count > 350 cells/mm3
    * Undetectable viral load
    * Maintained on modern therapeutic regimens utilizing non-cytochrome P450 (CYP)-interactive agents
    * No history of AIDS-defining opportunistic infections
15. Subject is known to be positive for hepatitis B or C infection, with the exception of those with an undetectable viral load within 3 months (Hepatitis B or C testing is not required for eligibility assessment).
16. Known hepatic cirrhosis or severe preexisting hepatic impairment.
17. Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to known cardiopulmonary disease defined as unstable angina, clinically significant arrhythmia, congestive heart failure (New York Heart Association Class III or IV; see Appendix 7), and/or ST elevation myocardial infarction within 6 months before first dose, or severe symptomatic pulmonary hypertension requiring pharmacologic therapy, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. As an example, well-controlled atrial fibrillation would not be an exclusion whereas uncontrolled atrial fibrillation would be an exclusion. Patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled.
18. Subject has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study.
19. Treatment with strong Cytochrome P450, family 3, subfamily A (CYP3A) inducers (see Appendix 8) within 14 days before the first dose of pevonedistat.
20. Patients with uncontrolled coagulopathy or bleeding disorder.
21. High blood pressure which cannot be controlled by standard treatments
22. Prolonged rate corrected QT (QTc) interval ≥ 500 msec, calculated according to institutional guidelines.
23. As infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control and no signs of systemic inflammatory response beyond low grade fever that makes patient clinically unstable in the opinion of the investigator. Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control.
24. Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent and until toxicity from this has resolved to grade 1 or less; if the half-life of the agent is unknown, patients must wait 4 weeks prior to first dose of study treatment.
25. Systemic antineoplastic therapy for malignant conditions other than myeloid neoplasms within 14 days before the first dose of any study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | through study completion, an average of 1 year
  Time from the date of randomization to the date of death.

SECONDARY OUTCOMES:
Event-free survival (EFS) | through study completion, an average of 1 year
  Time from randomization to the date of the occurrence of any of the following events: progressive disease, failure to achieve complete response or complete remission with incomplete blood count recovery at 6 months after initiation of treatment, relapse from complete response (CR)/ incomplete complete response (CRi) or death from any cause, whichever occurs first
Composite complete remission | through study completion, an average of 1 year
  The proportion of subjects with complete response plus complete remission with incomplete blood count recovery
Overall response rate | through study completion, an average of 1 year
  The proportion of subjects with complete response plus complete remission with incomplete blood count recovery plus partial response
Cumulative incidence of relapse | through study completion, an average of 1 year
  Calculated using the competing risk method (Fine & Gray)
Health status/quality of life | through study completion, an average of 1 year
  Global health status/quality of life based on patient reported outcome EORTC Quality of life questionnaire (QLQ)-C30 and supplemental items.
Health status/quality of life | through study completion, an average of 1 year
  Global health status/quality of life based on patient reported outcome: EQ-5D-5L questionnaire.
Use of medical resources determined by the use of antibiotics | through study completion, an average of 1 year
  Compare the use of antibiotics during the study between treatment groups
Use of medical resources determined by the use of transfusions | through study completion, an average of 1 year
  Compare the use of transfusions during the study between treatment groups
Use of medical resources determined by the number of hospital admissions | through study completion, an average of 1 year
  Compare the number of hospital admissions during the study between treatment groups
Pharmacokinetic | At day 1, 3 and 5 of cycle 1, cycle 2 and cycle 3 (each cycle is 28 days)
  Plasma concentration of Pevonedistat
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | through study completion (an average of 1 year)
  Adverse events of Pevonedistat plus Azacitidine versus Azacitidine regimen
Quality of composite complete remission determined by the minimal residual disease determined by RT-qPCR in the NPM1+ and CBF subsets and in bone marrow by MPFC in the remaining patients | through study completion, an average of 1 year
  To evaluate the quality of composite complete remission determining the minimal residual disease in patients with complete remission and complete remission with incomplete blood count recovery
Overall survival based on somatic mutations | through study completion, an average of 1 year
  To explore relationship of somatic mutations at baseline with overall survival
Event free survival based on somatic mutations | through study completion, an average of 1 year
  To explore relationship of somatic mutations at baseline with event free survival
Overall response rate based on somatic mutations | through study completion, an average of 1 year
  To explore relationship of somatic mutations at baseline with the overall response rate
Overall survival based on cytogenetic abnormalities | through study completion, an average of 1 year
  To explore relationship of cytogenetic abnormalities at baseline with overall survival
Event free survival based on cytogenetic abnormalities | through study completion, an average of 1 year
  To explore relationship of cytogenetic abnormalities at baseline event free survival
Overall response rate based on cytogenetic abnormalities | through study completion, an average of 1 year
  To explore relationship of cytogenetic abnormalities at baseline with the overall response rate
Red blood cells transfusion transfusion Independence (no use of red blood cells transfusion for a period of at least 8 weeks) | through study completion, an average of 1 year
  To determine if PEVO + AZA increase the duration of red blood cells transfusion Independence (transfusion independence requires that the patient receive no red blood cells transfusions for a period of at least 8 weeks)
Platelet transfusion Independence (no use of platelets transfusión for a period of at least 8 weeks) | through study completion, an average of 1 year
  To determine if PEVO + AZA increase the duration of platelets transfusion Independence (transfusion independence requires that the patient receive no platelets transfusions for a period of at least 8 weeks)
Biomarkers (CBF) predictive of PEVO activity | through study completion, an average of 1 year
  To assess biomarkers (CBF) predictive of PEVO activity evaluated by the overall response rate and minimal residual disease
Biomarkers (FLT3-ITD) predictive of PEVO activity | through study completion, an average of 1 year
  To assess biomarkers (FLT3-ITD) predictive of PEVO activity evaluated by the overall response rate and minimal residual disease
Biomarkers (NPM1) predictive of PEVO activity | through study completion, an average of 1 year
  To assess biomarkers (NPM1) predictive of PEVO activity evaluated by the overall response rate and minimal residual disease
Biomarkers (P53) predictive of PEVO activity | through study completion, an average of 1 year
  To assess biomarkers (P53) predictive of PEVO activity evaluated by the overall response rate and minimal residual disease
Biomarkers (IDH1/IDH2 ) predictive of PEVO activity | through study completion, an average of 1 year
  To assess biomarkers (IDH1/IDH2) predictive of PEVO activity evaluated by the overall response rate and minimal residual disease

CONTACTS AND LOCATIONS:
Locations (62):
- Spain (62):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Txagorritxu, Vitoria-Gasteiz, Alava
  - ICO Badalona- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO Hospitalet- Hospital Duran i Reynals, Hospitalet Del Llobregat, Barcelona
  - Hospital Universitario Donostia, San Sebastián, Guipuzcoa
  - Complejo Hospitalario de Jaén, Jaén, Jaen
  - Complejo Hospitalario Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Regional Universitario de Málaga, Málaga, Malaga
  - Hospital Universitario Virgen de la Victoria, Málaga, Malaga
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario Virgen del Rocío, Seville, Sevila
  - Hospital General Nuestra Señora del Prado, Talavera de la Reina, Toledo
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Hospital Universitario de Galdakao, Galdakao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Dr. José Molina Orosa, Arrecife
  - Hospital San Agustin, Avilés
  - Complejo Asistencial de Ávila, Ávila
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Vithas Xanit Internacional, Benalmádena
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Universitario de Castellón, Castelló
  - Complejo Hospitalario de Cáceres, Cáceres
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital General Universitario de Elche, Elche
  - ICO Girona- Hospital Universitari Dr Josep Trueta, Girona
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital San Jorge, Huesca
  - Complejo Hospitalario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Madrid Norte Sanchinarro, Madrid
  - Hospital Quirón de Málaga, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Son Llàtzer, Palma de Mallorca
  - Complexo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca
  - Complejo Hospitalario Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital General de Segovia, Segovia
  - Hospital de Valme, Seville
  - Hospital Universitari Joan XXIII, Tarragona
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset Aleixandre, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Background] Soucy TA, Smith PG, Milhollen MA, Berger AJ, Gavin JM, Adhikari S, Brownell JE, Burke KE, Cardin DP, Critchley S, Cullis CA, Doucette A, Garnsey JJ, Gaulin JL, Gershman RE, Lublinsky AR, McDonald A, Mizutani H, Narayanan U, Olhava EJ, Peluso S, Rezaei M, Sintchak MD, Talreja T, Thomas MP, Traore T, Vyskocil S, Weatherhead GS, Yu J, Zhang J, Dick LR, Claiborne CF, Rolfe M, Bolen JB, Langston SP. An inhibitor of NEDD8-activating enzyme as a new approach to treat cancer. Nature. 2009 Apr 9;458(7239):732-6. doi: 10.1038/nature07884. PMID 19360080
- [Background] Lin JJ, Milhollen MA, Smith PG, Narayanan U, Dutta A. NEDD8-targeting drug MLN4924 elicits DNA rereplication by stabilizing Cdt1 in S phase, triggering checkpoint activation, apoptosis, and senescence in cancer cells. Cancer Res. 2010 Dec 15;70(24):10310-20. doi: 10.1158/0008-5472.CAN-10-2062. PMID 21159650
- [Background] Milhollen MA, Narayanan U, Soucy TA, Veiby PO, Smith PG, Amidon B. Inhibition of NEDD8-activating enzyme induces rereplication and apoptosis in human tumor cells consistent with deregulating CDT1 turnover. Cancer Res. 2011 Apr 15;71(8):3042-51. doi: 10.1158/0008-5472.CAN-10-2122. Epub 2011 Apr 12. PMID 21487042
- [Result] Sarantopoulos J, Shapiro GI, Cohen RB, Clark JW, Kauh JS, Weiss GJ, Cleary JM, Mahalingam D, Pickard MD, Faessel HM, Berger AJ, Burke K, Mulligan G, Dezube BJ, Harvey RD. Phase I Study of the Investigational NEDD8-Activating Enzyme Inhibitor Pevonedistat (TAK-924/MLN4924) in Patients with Advanced Solid Tumors. Clin Cancer Res. 2016 Feb 15;22(4):847-57. doi: 10.1158/1078-0432.CCR-15-1338. Epub 2015 Sep 30. PMID 26423795
- [Result] Swords RT, Coutre S, Maris MB, Zeidner JF, Foran JM, Cruz J, Erba HP, Berdeja JG, Tam W, Vardhanabhuti S, Pawlikowska-Dobler I, Faessel HM, Dash AB, Sedarati F, Dezube BJ, Faller DV, Savona MR. Pevonedistat, a first-in-class NEDD8-activating enzyme inhibitor, combined with azacitidine in patients with AML. Blood. 2018 Mar 29;131(13):1415-1424. doi: 10.1182/blood-2017-09-805895. Epub 2018 Jan 18. PMID 29348128
- [Result] Dombret H, Seymour JF, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Bernal del Castillo T, Al-Ali HK, Martinelli G, Falantes J, Noppeney R, Stone RM, Minden MD, McIntyre H, Songer S, Lucy LM, Beach CL, Dohner H. International phase 3 study of azacitidine vs conventional care regimens in older patients with newly diagnosed AML with >30% blasts. Blood. 2015 Jul 16;126(3):291-9. doi: 10.1182/blood-2015-01-621664. Epub 2015 May 18. PMID 25987659
- [Result] Shah JJ, Jakubowiak AJ, O'Connor OA, Orlowski RZ, Harvey RD, Smith MR, Lebovic D, Diefenbach C, Kelly K, Hua Z, Berger AJ, Mulligan G, Faessel HM, Tirrell S, Dezube BJ, Lonial S. Phase I Study of the Novel Investigational NEDD8-Activating Enzyme Inhibitor Pevonedistat (MLN4924) in Patients with Relapsed/Refractory Multiple Myeloma or Lymphoma. Clin Cancer Res. 2016 Jan 1;22(1):34-43. doi: 10.1158/1078-0432.CCR-15-1237. Epub 2015 Nov 11. PMID 26561559
- [Result] Bhatia S, Pavlick AC, Boasberg P, Thompson JA, Mulligan G, Pickard MD, Faessel H, Dezube BJ, Hamid O. A phase I study of the investigational NEDD8-activating enzyme inhibitor pevonedistat (TAK-924/MLN4924) in patients with metastatic melanoma. Invest New Drugs. 2016 Aug;34(4):439-49. doi: 10.1007/s10637-016-0348-5. Epub 2016 Apr 8. PMID 27056178
- See also: Web page of the sponsor of the study — https://www.fundacionpethema.es